CLINICAL TRIAL: NCT00141531
Title: Phase II Study of Intravesical Instillation of EOQUIN™ in High Risk Superficial Bladder Cancer
Brief Title: Phase II Trial of EOquin in High-risk Superficial Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPI 05-003; 503
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Bladder Neoplasms
Keywords: Bladder cancer; Superficial; Carcinoma in situ; Intravesical instillation; Chemotherapy; Adjuvant
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma in Situ | interventions — apaziquone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Apaziquone (Active Comparator)
  Interventions: Drug: Apaziquone

INTERVENTIONS:
Drug: Apaziquone — Apaziquone (EOquinTM) 4 mg/40 mL was administered by intravesical instillation once a week for 6 consecutive weeks.
  In addition, patients with CIS were to receive further maintenance therapy of 3 weekly apaziquone (EOquinTM) instillations at 3, 6, and 12 months from the date of histological diagnosis.
  Other Names: EOquin

SUMMARY:
A non-randomized, open-label phase II study to explore the feasibility, time to recurrence, duration of response and safety of the adjuvant intravesical instillation of EOquin (apaziquone) in patients with high-risk superficial bladder tumors, and the response and duration of response in patients with carcinoma in situ of the bladder.

DETAILED DESCRIPTION:
Endpoints: Time to recurrence, duration of response and safety

Number of Patients: 53 patients

Study Design: Non-randomized, open-label study.

Key Inclusion Criteria: High-risk patients according to EAU criteria defined as

* pT1 and/or Grade 2b-3, or multiple and highly recurrent
* histologically confirmed carcinoma in situ (CIS)

Key Exclusion Criteria:

pTa Grade 1 or pT1 Grade 1 tumors, existing urinary tract infection or recurrent severe bacterial cystitis; those who cannot tolerate intravesical administration or intravesical surgical manipulation due to the presence of concomitant serious illness; no prior intravesical chemotherapy or immunotherapy in the last three months; no prior EOquin treatment (intravenous or intravesical) in last 12 months.

Study Treatment:

All patients will receive intravesical instillation of EOquin™ 4-mg/40 mL instillate once a week for six consecutive weeks

Patient with carcinoma in situ (CIS) will receive further maintenance therapy with 3 consecutive weekly EOquin instillations at the following time points: 3, 6, 12, 18, and 24 months from the date of TUR. At 3-month follow up visit patients will undergo cystoscopic bladder biopsy and urine cytology. If bladder biopsy is negative at 3-month visit, the follow up during the remaining visits will be by cystoscopy and urine cytology only, which will be done prior to the start of maintenance therapy. In case of positive cytology presence of CIS has to be confirmed histologically with biopsies.

At 6 months follow-up, if biopsies are positive for CIS, no further maintenance therapy will be given; patient will be taken off-study.

Duration of Patient Participation:

Intravesical instillation of EOquin™ will be given once a week for six consecutive weeks. All patients will have follow-up evaluations carried out at 3, 6, 9, 12, 15 and 18 months from the TUR date or until progressive disease is observed. In case of recurrence, patients will go off the study and further treatment will be at the investigator's discretion.

Off Study:

Patients will be taken off the study:

* Upon first recurrence and or progression
* Persistent CIS at 6 months follow up
* Recurrent CIS after biopsy proven complete response

ELIGIBILITY:
Inclusion Criteria:

1. Patients with high risk superficial bladder cancer according to EAU criteria defined as:

* pT1 and/or Grade 2b-3, or multiple and highly recurrent
* histologically confirmed carcinoma in situ 2. All visible lesions must be completely removed by transurethral resection (TUR) at entry to the study 3. Normal bimanual examination under anesthesia (no palpable masses) 4. Absence of upper urinary tract tumor confirmed by intravenous pyelography (IVP) or CT scan or retrograde urogram within 6 months from the beginning of treatment 5. Patient with ZUBROD-ECOG-WHO performance status of 0-2 (see Appendix 2) 6. Over 18 years of age 7. Patients must be fully informed of the investigational nature of the study and signed written informed consent must be obtained prior to any study specific investigations.

Exclusion Criteria:

1. Patients having muscle-invasive disease (T2 or greater)
2. Prior intravesical treatment (chemotherapy or immunotherapy) within the last 3 months
3. Patients with existing urinary tract infection or recurrent severe bacterial cystitis
4. Patients with urogenital tumors with histology other than transitional cell carcinoma (i.e., squamous cell or adenocarcinoma) or with transitional carcinoma involving the upper tract or the prostatic urethra
5. Patients with history of other primary malignancy (other than squamous or basal cell skin cancers or cone biopsied Cis of the uterine cervix or prostate carcinoma treated curatively with normal PSA values at inclusion) in the last five years
6. Patients with active, uncontrolled impairment of the renal, hepatobiliary, cardiovascular, gastrointestinal, urogenital, neurologic or hematopoietic systems which, in the opinion of the investigator, would predispose to the development of complications from the administration of intravesical therapy and or general anesthesia
7. Patients who, in the opinion of the investigator, cannot tolerate intravesical administration or intravesical surgical manipulation (cystoscopy, biopsy) due to the presence of concomitant serious illness (i.e. uncontrolled cardiac or respiratory disorders)
8. Women who are pregnant or lactating. Individuals of reproductive potential may not participate unless agreeing to use an effective contraceptive method for themselves and/or their sexual partner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2005-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Time to progression / Duration of remission following transurethral resection of superficial bladder cancer | 18 months

SECONDARY OUTCOMES:
Additional safety data | 18 months
Rate of upstaging on recurrence | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Witjes, MD, Prof., Study Chair — Urology Division, St Radboud University Hospital, Nijmegen, the Netherlands; Kees Hendricksen, MD, Study Director — St Radboud University Hospital, Nijmegen, the Netherlands
Locations (1):
- St Radboud University Hospital, Nijmegen, Netherlands